# **Gut Microbiome and p-Inulin in Hemodialysis**

A multi-center study to characterize the gut microbiome of individuals with end-stage renal disease treated with maintenance hemodialysis, and to explore effects of p-inulin on the gut microbiome

**Funding Sponsor:** National Institutes of Diabetes and Digestive

and Kidney Diseases

National Institutes of Health

2 Democracy Plaza

6707 Democracy Boulevard Bethesda, MD 20892-5458

Protocol Number: NA

Initial version: V1.0, July 1, 2015

Amended: V2.0, September 9, 2015

Amended: [date]

# **Table of Contents**

| LI | ST OF AF | BREVIATIONS | IV |
|---|---|---|---|
| ST | UDY SU | MMARY | V |
| 1 | INTR | ODUCTION | 1 |
| | 1.1 | BACKGROUND | 1 |
| | 1.2 | STUDY AGENT | |
| | 1.3 | CLINICAL DATA ON PREBIOTICS AND P-INULIN | |
| | 1.4 | Dose Rationale and Risk/Benefits | |
| | 1.4.1 | Risks | 5 |
| 2 | STUI | DY OBJECTIVES | 5 |
| | 2.1 | PRIMARY OBJECTIVES | 5 |
| | 2.2 | SECONDARY OBJECTIVES | |
| _ | | | |
| 3 | | DY DESIGN | |
| | 3.1 | GENERAL DESIGN | |
| | 3.2 | STUDY ENDPOINTS | |
| | 3.2.1 | · | |
| | 3.2.2 | Secondary Endpoints | 6 |
| 4 | PAR | FICIPANT SELECTION AND WITHDRAWAL | 7 |
| | 4.1 | INCLUSION CRITERIA | 7 |
| | 4.2 | EXCLUSION CRITERIA | 7 |
| | 4.2.1 | Women of Childbearing Potential | 8 |
| | 4.3 | RECRUITMENT | |
| | 4.4 | EARLY WITHDRAWAL OF PARTICIPANTS AND EARLY STUDY TERMINATION | |
| | 4.4.1 | , · | |
| | 4.4.2 | Dose Reduction and Discontinuation of p-Inulin | 9 |
| 5 | STU | DY PROCEDURES | 9 |
| | 5.1 | STUDY VISIT SCHEDULE | 9 |
| | 5.1.1 | Pre-screening Activities | 10 |
| | 5.1.2 | Screening/Baseline Visit | 10 |
| | 5.1.3 | Week 4, 8, 12, 16, 20, 24, and 28 Visits and Weekly Telephone Contacts | 10 |
| | 5.2 | BIOSAMPLE COLLECTION PROCEDURES AND SCHEDULE | |
| | 5.2.1 | | _ |
| | 5.2.2 | | |
| | 5.2.3 | | |
| | 5.2.4 | | _ |
| | 5.2.5 | | |
| | 5.3 | STOOL AND BLOOD ANALYSES | |
| | 5.3.1 | , | |
| 6 | | DY AGENT | |
| | 6.1 | DESCRIPTION | |
| | 6.2 | TREATMENT REGIMEN | |
| | 6.3 | ADMINISTRATION OF STUDY AGENT | 16 |

| | 6.4 | RECEIVING, STORING, DISPENSING AND RETURNING STUDY AGENT | 16 |
|---|---|---|---|
| | 6.4.1 | | |
| | 6.4.2 | | |
| | 6.4.3 | | |
| | 6.4.4 | | |
| | 6.5 | PARTICIPANT ADHERENCE MONITORING | |
| | 6.6 | CONCOMITANT THERAPY | |
| _ | | | |
| 7 | | ISTICAL PLAN | |
| | 7.1 | Sample Size Determination | |
| | 7.2 | MISSING DATA | |
| | 7.3 | STATISTICAL METHODS | |
| | 7.3.1 | , | |
| | 7.3.2 | , , | |
| | 7.3.3 | , , , , , , , | |
| | 7.3.4 | • | |
| | 7.3.5 | Analysis of Safety | 21 |
| 8 | SAFE | TY AND ADVERSE EVENTS | 21 |
| | 8.1 | Definitions | 21 |
| | 8.1.1 | Adverse Event | 22 |
| | 8.1.2 | Serious Adverse Event | 22 |
| | 8.1.3 | Unanticipated Problems Involving Risk to Participants or Others | 22 |
| | 8.1.4 | · | |
| | 8.2 | ADVERSE EVENT REPORTING PERIOD | |
| | 8.2.1 | Post-study Adverse Event | 23 |
| | 8.3 | RECORDING OF ADVERSE EVENTS | |
| | 8.3.1 | Anticipated Adverse Events | 23 |
| | 8.4 | REPORTING OF SERIOUS ADVERSE EVENTS AND UNANTICIPATED PROBLEMS | |
| | 8.4.1 | | |
| | 8.4.2 | | |
| | 8.5 | MEDICAL MONITORING | |
| | 8.5.1 | Independent Data and Safety Monitoring Board (DSMB) | 26 |
| 9 | DAT | A MANAGEMENT | 26 |
| פ | | | |
| | 9.1 | DATA QUALITY | |
| | 9.1.1 | • , | |
| | 9.1.2 | , | |
| | 9.2 | DATA SECURITY | |
| | 9.2.1 | , | |
| | 9.3 | Source Documents | |
| | 9.3.1 | • | |
| | 9.3.2 | 3 , , , | |
| | 9.3.3 | 9 | |
| | 9.3.4 | Records Retention | 29 |
| 10 | STUE | PY MONITORING, AUDITING, AND INSPECTING | 29 |
| | 10.1 | Study Monitoring Plan | |
| | 10.2 | Auditing and Inspecting | 20 |

| 11 E | ETHICAL CONSIDERATIONS | 30 |
|------|------------------------------------|----|
| 12 S | STUDY FINANCES | 30 |
| 12.1 | 1 Funding Source | 30 |
| 12.2 | 2 CONFLICT OF INTEREST | 30 |
| 12.3 | 3 PARTICIPANT STIPENDS OR PAYMENTS | 30 |
| 13 P | PUBLICATION PLAN | 30 |
| 14 R | REFERENCES | 32 |
| 15 A | ATTACHMENTS | 36 |
| 15.1 | 1 Study Procedures | 37 |
| 15.2 | 2 DSMB Charter | 38 |

#### **List of Abbreviations**

AE adverse event

CKD chronic kidney disease CRF case report form

CVD cardiovascular disease
DCC Data Coordinating Center
DMS data management system

DSMB Data and Safety Monitoring Board

ESRD end stage renal disease FOS fructo-oligosaccharides FTP File Transfer Protocol

HD hemodialysis

HIPAA Health Insurance Portability and Accounting Act

IDS Investigational Drug Service
IRB Institutional Review Board
MOP Manual of Procedures

NIDDK National Institute of Diabetes and Digestive and Kidney Diseases

NIH National Institutes of Health

OHRP Office of Human Research Protections

OTU operational taxonomic unit PHI protected health information

SAE serious adverse event
SAP statistical analysis plan
UAE unanticipated adverse event

# **Study Summary**

| Title | Gut Microbiome and p-Inulin in Hemodialysis |
|---|---|
| Short Title | Gut Microbiome in HD |
| Protocol Number | NA |
| Phase | Phase I |
| Methodology | Non-randomized, open label, 3-period crossover trial, with repeated measures within period |
| Study Duration | 28 weeks for participant; 15 months for full study (projected) |
| Study Center(s) | Brigham and Women's Hospital |
| | George Washington University |
| | University of Washington |
| | Vanderbilt University |
| | University of Pennsylvania (Data Coordinating Center) |
| Objectives | To evaluate intra- and inter-participant variability in the composition and metabolic products of the gut microbiome |
| | To evaluate the tolerability and short-term safety of p-inulin |
| | To assess the feasibility of sample collection in this population |
| Number of Participants | Up to 20 individuals will be enrolled until 10 participants complete the first 20 weeks of |
| | the study with satisfactory completeness of biosample collection |
| Diagnosis and Main<br>Inclusion Criteria | End-stage renal disease; treatment with maintenance hemodialysis |
| Study Product, Dose,<br>Route | p-Inulin 8 g twice daily, administered orally |
| Duration of administration | 12 weeks |
| Major Outcomes | Intra-participant variability in the gut microbiome composition |
| | Intra-participant variability in the metabolic products of the gut microbiome |
| | Tolerability of p-inulin |
| Statistical Methodology | Alpha-diversity of bacterial genera will be derived at each time point, and intra-class correlation coefficients, using mixed models, will be estimated to evaluate diversity of multiple observations within each individual |
| | UniFrac distances will be derived as beta diversity measures of inter-participant variability to characterize the compositional dissimilarity of the microbiome between two individuals |
| | A repeated measures MANOVA of UniFrac distances will be used to assess the |
| | changes of the overall microbial compositions over time. |
| | <ul> <li>Longitudinal mixed-effect models will be applied to study change of metabolites<br/>before and after p-inulin treatment, and to identify the metabolites that change<br/>after p-inulin treatment</li> </ul> |
| | Longitudinal analyses of metabolites, with time-varying covariates (microbiome diversity or microbial genera) will be conducted to identify the microbial genera associated with changes of metabolites due to p-inulin treatment |

### 1 Introduction

This document is a protocol for a human research study. This study is to be conducted according to US and international standards of Good Clinical Practice, applicable government regulations, and the research policies and procedures in effect at the institutions where the study is implemented.

### 1.1 Background

A substantial body of work implicates inflammation as an important contributor to the morbidity and mortality associated with end-stage renal disease (ESRD) and, in particular, to accelerated cardiovascular disease. However, the etiology of unprovoked inflammation in ESRD is not well understood. Proposed etiological factors include chronic sub-clinical infections, volume overload, oxidative stress, sympathetic activation, malnutrition, and vitamin D deficiency. Alterations in the intestinal microbiome (dysbiosis) are increasingly recognized as potential causes of inflammation in ESRD patients. <sup>8-12</sup>

The human gut harbors ~10<sup>14</sup> bacteria, and the metabolic potential of the gut microbiota is enormous. <sup>15</sup> Intestinal bacteria perform a multitude of functions, and the microbial flora can be considered a metabolically active endogenous "organ." Under physiological conditions, the microbiota provide complementary functions by participating in metabolic activities that are not fully evolved in the human host such as break down of non-digestible plant polysaccharides, <sup>16</sup> synthesis of certain vitamins, <sup>17</sup> biotransformation of conjugated bile acids <sup>18</sup> and degradation of dietary oxalates. <sup>19</sup> Additionally, postnatal colonization of the intestine educates the immune system and reduces allergic responses to food and environmental antigens. <sup>20</sup>

Alterations in the gut microbiome have been demonstrated in patients with ESRD. 9,12 Individuals with uremia have greatly increased counts of both aerobic (~10<sup>6</sup> bacteria/ml) and anaerobic (~10<sup>7</sup> bacteria/ml) organisms in the duodenum and jejunum.<sup>21</sup> The microbial flora of the lower intestinal tract has also been shown to be altered in patients with non-dialysis dependent chronic kidney disease. The most notable changes are reductions in both the Lactobacillaceae and Prevotellaceae families. <sup>9</sup> Hida et al. studied the colonic composition of microbiota in healthy controls and hemodialysis patients.<sup>22</sup> The number of aerobic bacteria such as Enterobacteria and Enterococci was found to be approximately 100 times higher in patients treated with maintenance hemodialysis than in controls. Among anaerobic bacteria, hemodialysis patients had significantly lower organism counts for Bifidobacteria and higher organism counts for Clostridium perfringens.<sup>22</sup> Vaziri et al. showed significant differences in the abundance of 190 microbial operational taxonomic units (OTUs) between the ESRD and the normal control individuals. <sup>9</sup> In order to isolate the effect of kidney failure, the investigators examined the gut microbiota in nephrectomized rats. <sup>9</sup> The study revealed substantially lower "species richness" as measured by the number of OTUs in the nephrectomized rats compared to the controls. The intestinal dysbiosis may be a direct or indirect effect of uremia.<sup>23,24</sup> For example, loss of kidney function leads to secretion of urea into the gastrointestinal tract. Hydrolysis of urea by bacterial urease generates large quantities of ammonia which alters the growth of commensal bacteria. 23,24 Other contributing indirect factors relevant to patients with kidney failure include decreased consumption of dietary fiber, 25-27

frequent use of antibiotics,<sup>28,29</sup> slow colonic transit,<sup>30,31</sup> metabolic acidosis,<sup>32,33</sup> intestinal wall edema,<sup>34-36</sup> and possibly oral iron intake.<sup>37,38</sup>

There are multiple mechanisms by which such alterations in the gut microbiota might contribute to ESRD-associated inflammation and cardiovascular disease including 1) increased production of bacteria-derived solutes (e.g., p-cresol or p-cresyl sulfate) that are retained in kidney failure, <sup>39-41</sup> and 2) increased translocation into the circulation of bacterial-derived endotoxin across an impaired intestinal barrier. <sup>10,11,42,43</sup> Elevated serum concentrations of total and free p-cresol are associated with cardiovascular events and mortality among patients treated with maintenance hemodialysis, <sup>44,45</sup> and experimental as well as clinical studies indicate that endotoxin is involved in multiple steps of atherogenesis. <sup>46,47</sup> Endotoxin provokes a host of responses by binding to the CD14 receptor. <sup>48</sup> Elevation in the concentration of soluble CD14 (sCD14), an indicator of CD14 receptor activation, is an independent predictor of mortality among patients treated with maintenance hemodialysis. <sup>10,11</sup>

Prebiotics are microbial feed supplements that beneficially affect the host by improving its intestinal microbial balance and re-establishing symbiosis. Treatment with the prebiotic p-inulin increases intestinal growth of beneficial bacteria such as bifidobacteria. Increases in bifidobacteria are associated with attenuation of inflammation and improvement in intestinal barrier function. Other reported effects of prebiotic supplementation include optimizing the immune response, decreasing endotoxin generation, and enhancing metabolic capabilities. Preliminary evidence indicates that prebiotics are effective in reducing the plasma concentration of p-cresyl sulfate in hemodialysis patients. In a single center, non-randomized, open-label phase I/II study of hemodialysis patients, treatment with p-inulin for 4 weeks was accompanied by a reduction in the p-cresyl sulfate generation rate and a 20% decrease in its serum concentration.

There are important potential benefits of intervening to restore symbiosis to the gut microbiota in patients with ESRD. However, before conducting clinical trials of such interventions, important gaps must be filled in the understanding of the composition, function and stability of the gut microbiota in patients with ESRD. The purpose of the Microbiome and P-Inulin in Hemodialysis Study is to fill some of these gaps in anticipation of ultimately investigating the therapeutic potential of altering the composition and/or function of the gut microbiome in this patient population. Intensive biosample collection from a small number of patients treated with hemodialysis before, during, and after treatment with p-inulin will be performed in order to generate information about within-participant and between-participant variability in the composition and metabolic products of the gut microbiome. The study will also provide information about the tolerability and safety of p-inulin and the feasibility of biosample collection.

# 1.2 Study Agent

p-Inulin (oligofructose-enriched inulin) is a prebiotic. Inulin-type prebiotics are members of a larger group of compounds called "fructans," which encompasses all naturally occurring plant oligo- and polysaccharides in which one or more fructosyl-fructose linkages comprise the majority of glycosidic bonds. Inulin is present in vegetables with high fiber content such as sugar beets, leeks, onions, garlic and

asparagus. The basic inulin, derived from chicory root, is treated with specific bacterial enzymes that break down the long chain inulin to the short chain oligofructose in 95% pure form. Short-chain oligofructose is mixed with inulin in equal parts to prepare the final product, p-inulin.<sup>59</sup> This composition allows the short chain oligofructose to be fermented in the proximal (right) colon and the long chain molecule, inulin, to be fermented in the distal colon.<sup>60</sup> The end products of fermentation are gases (such as carbon dioxide and hydrogen), lactate, and short-chain fatty acids.

Preliminary evidence in individuals with preserved kidney function indicates that p-inulin promotes growth of bifidobacteria, reduces endotoxin generation, attenuates inflammation, decreases generation of uremic toxins and improves metabolic function. 12,49,61,62

Inulin-type prebiotics received the designation of "generally recognized as safe" in 1992.<sup>63</sup>

### 1.3 Clinical Data on Prebiotics and p-Inulin

A large number of studies have been performed examining the effect of prebiotics in a variety of conditions including obesity,  $^{64,65}$  HIV infection  $^{66,67}$  and gastrointestinal diseases. Bouhnik et al. showed that four weeks of treatment with short-chain fructo-oligosaccharides increases fecal bifidobacteria counts. In a small, randomized double-blind, placebo-controlled trial, 31 participants who had received radiotherapy were randomized either to p-inulin or maltodextrin-containing placebo for 4 weeks. Lactobacillus and bifidobacterium counts decreased with radiotherapy and recovered in the active treatment group but not in the placebo group. In another study, 49 individuals with diabetes were randomized to treatment with either inulin 10 g/day or a maltodextrin-containing placebo for 8 weeks. In comparison with placebo, inulin treatment improved insulin resistance and reduced plasma levels of lipopolysaccharide, hs-CRP and TNF- $\alpha$ .

There are a limited number of studies of prebiotic treatments in patients with ESRD (**Table 1**). In a pilot study of 22 patients receiving maintenance hemodialysis, treatment with 20 g of p-inulin for 4 weeks reduced the generation and serum concentration of p-cresol.<sup>58</sup> The authors reported that p-inulin was well tolerated and that there was excellent adherence with treatment. Nakabayashi showed that symbiotic treatment (Lactobacillus casei Shirota strain and Bifidobacterium breve Yakult strain as probiotics and galacto- ligosaccharides as prebiotics) three times per day for 2 weeks reduced p-cresol levels in maintenance hemodialysis.<sup>57</sup>

Table 1: Effect of pro-prebiotic on uremic toxins and inflammation

| Reference | Patient type (n) | Intervention | Comments |
|---|---|---|---|
| De Preter et al. <sup>72</sup> | Healthy participants (50) | Oligofructose-enriched | ↓ Urinary excretion of p-cresol |
| | | inulin | |
| Dewulf et al. <sup>64</sup> | Obese women (30) | Inulin/oligofructose | ↓Endotoxemia |
| Schiffrin et al. <sup>73</sup> | Elderly participants (74) | Oligosaccharides | ↓TNF-alpha mRNA and IL-6 |
| | | | mRNA |
| | | | ↓Serum sCD14 |
| Kotzampassi et al. <sup>74</sup> | Trauma patients (65) | Probiotics along with | ↓ Rate of systemic |
| | | inulin, oat bran, pectin, | inflammatory response, |
| | | and resistant starch | syndrome, infections, severe |
| | | | sepsis, and mortality |
| Meijers et al. <sup>58</sup> | Hemodialysis patients (22) | Oligofructose-enriched | ↓ Serum p-cresyl sulfate and |
| | | inulin | generation rate |
| Nakabayashi et al. <sup>57</sup> | Hemodialysis patients (7) | Galacto-oligosaccharides | ↓ Serum p-cresol |
| | | and <i>L. casei</i> , and <i>B.</i> | |
| | | breve | |

#### 1.4 Dose Rationale and Risk/Benefits

A dose-dependent bifidogenic effect has been observed with p-inulin.  $^{49,75}$  Bouhnik et al. examined the dose dependent effect of 8 weeks treatment with short-chain fructo-oligosaccharides (SC-FOS).<sup>62</sup> Forty healthy volunteers were randomized to one of five groups: G<sub>0</sub> group (SC-FOS 0 g and saccharose 20 g) used as placebo; G<sub>2.5</sub> group (SC-FOS 2.5 g and saccharose 17.5 g); G5 group (SC-FOS 5 g and saccharose 15 g); G<sub>10</sub> group (SC-FOS 10 g and saccharose 10 g); and G<sub>20</sub> group (SC-FOS 20 g and saccharose 0 g). Bifidobacteria counts at Day 8 were greater in groups  $G_{10}$  and  $G_{20}$  compared with  $G_0$  and  $G_{2.5}$ . Total anaerobes increased at the 10 g daily dose, but not at lower doses, while no significant differences were found for Bacteroides, Lactobacillus, or Enterobacteriaceae. Excess flatus was significantly more frequent in participants consuming G<sub>20</sub>. The authors concluded that for healthy individuals consuming their usual diets, 10 g/day is the optimal dose in terms of tolerability and efficacy with respect to increasing fecal bifidobacteria. Gibson et al. reported that FOS at 15 g/day in three divided doses increased the proportion of Bifidobacteria from 6% to 22% in healthy adults during two weeks of use. The effect on Bifidobacteria was accompanied by significant decreases in Bacteroides, Clostridia, and Fusobacteria.<sup>49</sup> Meijers et al. showed that a dose of 20 g/day is tolerated by patients with ESRD; however, reports of abdominal symptoms were frequent.<sup>77</sup> Thus, the doses of 10 g and 20 g daily resulted in significant increases in fecal Bifidobacteria compared to lower doses, but with more abdominal symptoms at the higher dose. 49,59,76,78

In the current study, all participants will receive p-inulin at a dose of 8 g two times per day for a total daily dose of 16 g. Based on experience in non-ESRD populations, it is anticipated that this dose will have acceptable tolerability and sufficient efficacy. <sup>49, 62</sup>

#### 1.4.1 Risks

The most common side effects of p-inulin include gastrointestinal symptoms such as flatulence, bloating, abdominal distension, loose stools, and increased stool frequency.<sup>42</sup> These symptoms have been more frequently reported with inulin doses in the range of 15 to 30 g per day than with lower doses.<sup>79,80</sup> Gastrointestinal symptoms will be ascertained in this study using the Gastrointestinal Symptom Rating Scale.<sup>81</sup> Detailed collection of gastrointestinal symptoms is important for this population because these symptoms, particularly constipation, occur frequently in ESRD patients in the absence of p-inulin treatment. Participants are not expected to benefit from participating in this study. The data obtained from this study will be used to inform the design of a larger, placebo-controlled study to assess the therapeutic potential of altering the gut microbiome with p-inulin in hemodialysis patients.

# 2 Study Objectives

The overarching hypothesis motivating this exploratory study of variability of the human gut microbiome is that treatment with oligofructose enriched inulin (p-inulin) will alter the composition and/or function of the gut microbiome, and thereby reduce the generation of gut-derived uremic toxins, improve gut barrier function and attenuate systemic inflammation in patients treated with maintenance hemodialysis. In order to design a future clinical trial to test this hypothesis, information is needed about the following parameters from individuals receiving maintenance hemodialysis:

- 1) Intra-participant and inter-participant variability in the metabolic products and composition of the gut microbiome
- 2) Impact of p-inulin on the metabolic products and composition of the gut microbiome
- 3) Tolerability of p-inulin
- 4) Safety of p-inulin
- 5) Feasibility of collecting stool samples in this patient population

### 2.1 Primary Objectives

- To evaluate the within-participant variability of gut bacteria-derived metabolites and gut bacterial composition over an 8-week period during which there is no protocol-driven treatment
- To evaluate, using each participant as his/her own control, whether treatment with p-inulin for 12 weeks alters gut bacteria-derived metabolites and gut bacterial composition

### 2.2 Secondary Objectives

- To evaluate, using each participant as his/her own control, whether p-inulin alters levels of selected circulating inflammatory markers and mediators
- To assess between-participant variability of gut bacteria-derived metabolites and gut bacterial composition over an 8-week period during which there is no protocol-driven treatment
- To assess between-participant variability of gut bacteria-derived metabolites and gut bacterial composition during a 12-week period of treatment with p-inulin
- To evaluate the tolerability of p-inulin administered at a total daily dose of 16 g
- To evaluate the short-term safety of p-inulin administered at a total daily dose of 16 g
- To assess adherence to p-inulin treatment

- To explore the willingness of hemodialysis patients to enroll in a study requiring repeated collection of stool samples
- To explore participant adherence to the stool sample collection requirements
- To identify barriers to adhering to stool sample collection

# 3 Study Design

## 3.1 General Design

This is a non-randomized, open-label, crossover study. Participants will be followed during 3 sequential phases: 1) no intervention (8 week observational period), 2) p-inulin administration (12 week treatment period), and 3) no intervention (8 week observational period). The visit and stool and blood collection schedule for each phase is depicted in **Figure 1** and a detailed table of study procedures is provided in **Section 15.1**. Study participants will be recruited from four sites in the U.S.

**Baseline Visit** Week 4 Visit Week 8 Visit Week 12 Visit Week 16 Visit Week 20 Visit Week 24 Visit Week 28 Visit Medication, Screening/ ledication and Medication and Nedication and Enrollment/ Clinical Event Clinical Event Clinical Event. Clinical Event Clinical Event. Clinical Event Clinical Event and Tolerability Baseline Data Collection Dispense p-Inulin Review Review Review ال Weeks 10-19 Week 20 Week 21 . Weeks 21-28 Weeks 1-7 Week 8 Stool collection 2X per week 1X per week 2X per week 1X per week 2X per week 2X per week 1X per week Blood collection 1X per week 1X per week 1X per week 1X per week 1X per week 1X per week 1X per week Study Observation Completion Stop p-Inulin treatment Initiate p-Inulin treatment treatment and resume

no treatment

Figure 1. Visit and Biosample Collection Schedule

# 3.2 Study Endpoints

## 3.2.1 Primary Endpoints

Microbiome Characterization primary endpoints include:

- Within-participant variability in the metabolomic profile and targeted metabolites / inflammatory markers during the no treatment phases
- 2. Within-participant variability in the metabolomic profile and targeted metabolites / inflammatory markers during the p-inulin treatment phase

### 3.2.2 Secondary Endpoints

Microbiome Characterization secondary endpoints include:

 Within-participant change in the metabolomic profile and targeted metabolites / inflammatory markers after p-inulin treatment compared with pre-treatment

- 2. Within-participant variability in the bacterial composition of the stool during the no treatment phase
- 3. Within-participant variability in the bacterial composition of the stool during the p-inulin treatment phase
- 4. Within-participant change in the bacterial composition of the stool after p-inulin treatment compared with pre-treatment
- 5. Differences in the above measures between diabetic and non-diabetic participants
- 6. Within-study cohort variability in the metabolomic profile and targeted metabolites / inflammatory markers during the no treatment phase
- 7. Within-study cohort variability in the metabolomic profile and targeted metabolites / inflammatory markers during the p-inulin treatment phase
- 8. Within-study cohort change in the metabolomic profile and targeted metabolites / inflammatory markers after p-inulin treatment compared with pre-treatment

## Tolerability and Safety endpoints include:

- 1. Gastrointestinal symptoms
- 2. Early discontinuation of p-inulin
- 3. Reduction in p-inulin dose
- 4. Adverse events

### Study Feasibility endpoints include:

- 1. Enrollment refusal rate
- 2. Proportion of completed protocol-specified stool sample collections
- 3. Proportion of completed blood sample collections
- 4. Adherence to p-inulin assessed by packet counts
- 5. Participant withdrawal during each phase of the study

# 4 Participant Selection and Withdrawal

### 4.1 Inclusion Criteria

- a) Maintenance hemodialysis therapy for end-stage renal disease
- b) Age ≥ 18 years
- c) ≥90 days since hemodialysis initiation
- d) Self-reported average stool frequency of at least 1 every other day
- e) For women of childbearing potential, willingness to use a highly effective method of birth control for up to 4 weeks after the last dose of p-inulin. See **Section 4.2.1** for definition of childbearing potential and acceptable methods of birth control.
- f) Ability to provide informed consent

## 4.2 Exclusion Criteria

a) Use of prebiotics or probiotics during the past 8 weeks

- b) Consumption of probiotic yogurt during the past 2 weeks
- c) Use of antibiotics within the past 8 weeks
- d) Presence of HIV infection, chronic wound infection, osteomyelitis, or current hemodialysis vascular access infection
- e) Inflammatory bowel disease, chronic diarrhea, current C. difficile infection
- f) Cirrhosis or chronic active hepatitis
- g) Anticipated kidney transplantation, change to peritoneal dialysis, or transfer to another dialysis unit within 9 months
- h) Expected survival less than 9 months
- i) Pregnancy, anticipated pregnancy, or breastfeeding
- j) Incarceration
- k) Participation in another intervention study
- Severe anemia defined as hemoglobin <9.0 g/dl within the past 4 weeks as documented in the dialysis unit patient record

## 4.2.1 Women of Childbearing Potential

Women of childbearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Postmenopausal is defined as:

- Amenorrhea for ≥12 consecutive months without another cause or
- Women with irregular menstrual periods and a documented serum follicle stimulating hormone
   (FSH) level > 35 mIU/mL or
- Women on hormone replacement therapy (HRT)

Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or who are practicing abstinence, or have a partner who is sterile (e.g., vasectomy) should be considered to be of childbearing potential.

Acceptable methods of highly effective birth control include:

- Condom with spermicide
- Diaphragm and spermicide
- Cervical cap and spermicide
- Hormonal contraception

#### 4.3 Recruitment

Participants will be recruited from four Clinical Centers with a general goal of enrolling 3-5 participants at each site. Participants at dialysis units affiliated with investigator and co-investigator practices will be screened for eligibility. In addition to active screening of dialysis unit patient rosters by study personnel, informational handouts and brochures may be disseminated at affiliated dialysis units to allow potential participants to learn about the study and to contact investigators if interested. All study

materials must be approved by local Institutional Review Boards (IRB) before dissemination to potential study participants.

Dialysis unit laboratory studies, medical records at the investigator's institution, and treatment or medical history records at the dialysis unit will be reviewed to assess eligibility for enrollment. No study-specific testing is required to confirm eligibility, other than a serum pregnancy test for women of childbearing potential. Before approaching potential participants, the treating nephrologist will be contacted to assess suitability for enrollment.

Once preliminary eligibility is confirmed, written informed consent will be obtained by a qualified investigator or study site designee during an in-person visit. This visit may take place either at the local dialysis unit or at the investigator's institution in accordance with investigator and participant preferences.

Recruitment will continue until a total of 10 participants have satisfactorily completed the first 20 weeks of the study protocol.

Participants will be compensated for providing stool samples. Each Clinical Center is responsible for developing a compensation plan and schedule, and distributing payment.

### 4.4 Early Withdrawal of Participants and Early Study Termination

#### 4.4.1 Early Withdrawal of Participants

Reasons for premature withdrawal include pregnancy, death, and withdrawal of consent. Participants who are not able or willing to continue taking the study agent will be encouraged to remain in the study and continue biosample collection.

#### 4.4.2 Dose Reduction and Discontinuation of p-Inulin

Participants who are unable to tolerate p-inulin at a total dose of 16 g per day (8 g twice daily) will have the dose reduced to a total dose of 8 g per day (4 g twice daily). If the participant is unable to tolerate a total daily dose of 8 g, p-inulin will be discontinued.

If p-inulin is discontinued, study visits, sample collection and other procedures will continue as planned unless the participant withdraws consent for follow-up.

Participants who have reduction in dose or discontinuation of p-inulin because of intolerance are permitted, at the discretion of the site investigator, to resume taking p-inulin within the 12-week dosing phase.

# 5 Study Procedures

### 5.1 Study Visit Schedule

A schedule of study visits and procedures is provided in the Study Procedures Table in Section 15.1.

### **5.1.1** Pre-screening Activities

Patients at dialysis units affiliated with investigator and co-investigator practices will be screened for eligibility. Clinical Center study personnel will review dialysis unit records and other medical records to assess eligibility. The treating nephrologist for a potentially eligible patient will be contacted to further assess eligibility and obtain permission to contact the patient.

### 5.1.2 Screening/Baseline Visit

Patients who appear eligible based on pre-screening will be approached in person to determine interest in participation and confirm eligibility. Study personnel will discuss the study goals and procedures with the potential participant in detail. If the patient agrees to participate in the study, study personnel will review and assess understanding of the entire informed consent form before obtaining written informed consent from the participant. The consenting process will be performed by a qualified investigator or study site designee. Informed consent will be obtained and documented before any study procedures are performed.

The screening and baseline activities may take place over a single or multiple visits.

### **Screening/Baseline Visit Activities**

- Informed consent process
- Collection of baseline data including demographics, medical history, and medication use
  including recent and current use of prescription products, over-the-counter products, herbal
  supplements, vitamins, and prebiotic and probiotic use in any form. In addition, medical records
  from the dialysis facility will be reviewed to capture any non-reported data on recent
  medication use.
- Determination of eligibility
- Blood draw for baseline measurements (13 mL); blood draw must be performed before the start of the dialysis session
- Blood draw for serum pregnancy test for women of childbearing potential
- Instruction in stool sample collection and storage
- Dietary assessment using food frequency questionnaire
- Gastrointestinal symptom assessment questionnaire

Enrolled participants will be instructed not to change their dietary patterns, if possible, during the study.

See Section 5.2 for details regarding the blood and stool sample collection schedule.

### 5.1.3 Week 4, 8, 12, 16, 20, 24, and 28 Visits and Weekly Telephone Contacts

Participants will have in-person study visits at Weeks 4, 8, 12, 16, 20, 24 and 28. At each study visit, participants will be asked about emergency room visits, hospital admissions or any significant clinical events that occurred since the last visit. On a weekly basis, participants will be queried on antibiotic use in the previous week, and dialysis records will be reviewed for antibiotics administered at the dialysis unit. During the dosing phase, participants will also be asked questions to assess adherence with p-inulin.

Dietary assessment using the Block Food Frequency Questionnaire (<a href="https://nutritionquest.com">https://nutritionquest.com</a>) will be administered at Baseline and Weeks 8 (end of pre-treatment phase), 20 (end of treatment phase), and 28 (end of post-treatment phase).

#### Week 4 Visit

- Information on clinical events and current use of medications will be collected.
- Gastrointestinal symptom assessment questionnaire will be administered.

### Week 8 Visit

- Information on clinical events and current use of medications will be collected.
- Gastrointestinal symptom assessment questionnaire will be administered.
- Dietary assessment using a food frequency questionnaire will be administered to assess dietary patterns before starting p-inulin.
- A four week supply of p-inulin will be dispensed to the participant along with instructions for its use.
- To assess adherence to the study protocol, participants will be instructed to keep all unused study agent packets and bring them to the Week 12 visit.

### Week 12 Visit

- Information on clinical events and current medication use will be collected.
- Gastrointestinal symptom assessment questionnaire will be administered.
- Tolerability of p-inulin will be assessed by participant self-report. If participant has not been able to tolerate 16 g total daily dose, the dose may be reduced to a total daily dose of 8 g.
- Study personnel will collect, count and record the number of unused p-inulin packets.
- A four week supply of p-inulin will be dispensed.
- To assess adherence to the p-inulin treatment schedule, participants will be instructed to keep all unused study agent packets and bring them to the Week 16 visit.

#### Week 16 Visit

- Information on clinical events and current medication use will be collected.
- Gastrointestinal symptom assessment questionnaire will be administered.
- Tolerability of p-inulin will be assessed by participant self-report. If participant has not been able to tolerate 16 g total daily dose, the dose may be reduced to a total daily dose of 8 g.
- Study personnel will collect, count and record the number of unused p-inulin packets.
- A four week supply of p-inulin will be dispensed.
- To assess adherence to the p-inulin treatment schedule, participants will be instructed to keep all unused study agent packets and bring them to the Week 20 visit.

### Week 20 Visit

- Information on clinical events and current medication use will be collected.
- Gastrointestinal symptom assessment questionnaire will be administered.

- Dietary assessment using a food frequency questionnaire will be administered to assess dietary patterns during the p-inulin treatment period.
- Tolerability of p-inulin will be assessed. Study personnel will collect, count and record the number of unused p-inulin packets.

#### Week 24 Visit

- Information on clinical events and current medication use will be collected.
- Gastrointestinal symptom assessment questionnaire will be administered.

### Week 28 Visit (Study Completion)

- Information on clinical events and current medication use will be collected.
- Gastrointestinal symptom assessment questionnaire will be administered.
- Dietary assessment using a food frequency questionnaire will be administered to assess dietary patterns during the p-inulin treatment period.

# 5.2 Biosample Collection Procedures and Schedule

Stool samples will be collected at baseline, once weekly during weeks 1–7, 10–18 and 21-28, and twice weekly during weeks 8, 9, 19, and 20. The sample collection during weeks 21-28 (after p-inulin treatment) will allow detection of delayed alterations in response to p-inulin and will provide information about the durability of p-inulin effects.

Stool specimens will be obtained by study participants. Participants will be provided a commercial "toilet hat" stool specimen collection kit (specimen container, shipping box, Styrofoam cooler, and cold packs; Fisherbrand Commode Specimen Collection System; Thermo Fisher Scientific, Waltham, MA, USA), sample aliquot tubes, and gloves at the Baseline visit and as needed for resampling. Participants will be instructed on how to aliquot and store samples before bringing them to the research team.

Participants will bring the aliquoted stool samples on ice packs in the closed Styrofoam cooler to the clinical center or dialysis unit. Research staff will process samples according to Core Laboratory specifications and store at -80 °C for future shipment to the Core Laboratory. The aliquoting of samples is performed before freezing in order to minimize the number of freeze-thaw cycles. Detailed information regarding stool sample collection, storage, shipping, and participant training is provided in the Manual of Procedures (MOP).

Participants who do not provide the required number of stool samples will continue to be followed for the full duration of the study and will continue to be encouraged to provide samples in accordance with the protocol schedule.

All blood samples will be obtained on dialysis days before the start of the dialysis session and before any interaction between the blood and the dialyzer membrane. The volume of each sample will be 13 mL. Study staff will review the most recent hemoglobin lab results in the dialysis unit medical record. If this result is less than 9.0 g/dl, blood will not be collected until the hemoglobin value is 9.0 g/dl or greater.

Blood specimens will be processed and aliquoted according to the Core Laboratory specifications. Samples will be stored at -80° C for future shipment to the Core Laboratory. The MOP provides detailed information on blood specimen processing.

#### 5.2.1 Weeks 1-7

Stool and blood samples will be collected one time each week. Participants will be provided with written instructions about how to collect and store stool samples.

#### 5.2.2 Weeks 8-9

During the week before and the week after the change from no-treatment to p-inulin treatment, the frequency of stool sample collection will increase to two times per week. Blood collection will occur one time each week.

#### 5.2.3 Weeks 10-18

Stool and blood samples will be collected one time each week.

#### 5.2.4 Weeks 19-20

During the week before and the week after the change from p-inulin treatment to post-treatment, the frequency of stool sample collection will increase to two times per week. Blood collection will occur one time each week.

#### 5.2.5 Weeks 21-28

Stool and blood samples will be collected one time each week.

## 5.3 Stool and Blood Analyses

### 5.3.1 Metabolites and Inflammatory Markers.

Metabolites and inflammatory markers of interest that provide functional information about the gut microbiota or the host response are shown in **Table 2**. Both non-biased and targeted metabolomic profiling of the stool and blood will be performed. Inflammatory markers will be measured in the plasma samples.

Filtered fecal water or plasma samples will be used for the mass spectrometry-based metabolomic profiling. The process of metabolite extraction will include internal standards and follow standard protocols. The resulting extract will be divided into a liquid chromatography fraction and a gas chromatography fraction.

**Table 2. Stool and Blood Analytes of Interest** 

| | Stool | Blood |
|---------------------------------------------------------|-------|-------|
| Short chain fatty acids (butyrate, propionate, acetate) | + | + |
| Trimethylamine N oxide | + | + |
| Phenols | | |
| p-Cresyl sulfate | + | + |
| p-Cresyl glucuronide | + | + |
| Phenyl sulfate | + | + |
| Phenyl glucuronide | + | + |
| α-N-phenylacetyl-L-glutamine | + | + |
| Phenylpropionylglycine | + | + |
| Hippuric acid | + | + |
| 4-hydroxybenzoate | + | + |
| Phenylacetylglycine | + | + |
| Indoles | | |
| Indoxyl sulfate | + | + |
| Indoxyl glucuronide | + | |
| 5-hydroxyindole | + | |
| Indole-3-prioonic acid | + | |
| Indole-3-acetic acid | + | + |
| Polyamines | + | + |
| Metabolites of urea metabolism | + | + |
| Metabolites of creatinine metabolism | + | + |
| Allantoin | + | |
| Cytokines | | |
| IL-1β | | + |
| IL-2 | | + |
| IL-4 | | + |
| IL-6 | | + |
| IL-10 | | + |
| IL-17 | | + |
| IL-22 | | + |
| TNFα | | + |
| Endotoxin | | + |
| Myeloperoxdase (MPO) | | + |
| hsCRP | | + |
| HMGB1 | | + |
| TNF-R1 | | + |
| TNF-R2 | | + |
| Lipopolysaccharide binding protein (LBP) | | + |
| sCD14 | | + |

<u>Liquid chromatography/Mass spectrometry (LC/MS):</u> A 6590 Triple Quadrupole mass spectrometer (QQQ, Agilent Technologies, Santa Clara, CA) connected in the front end to Ultra Performance Liquid Chromatography will be used for Multiple Reaction Monitoring-based target metabolic quantification.1 Data acquisition in QQQ will be controlled using the Mass Hunter data acquisition software. Findings will be confirmed using selected reaction monitoring (SRM).

Gas chromatography/Mass spectroscopy (GC/MS): The derivatized samples will be injected into GC-MS, which is run using electron impact as the ionization source. Similar to the LC-based platform, detection of the metabolite would involve detection of its precursor followed by additional accurate mass detection of the product ions for the precursor by SRM. Each of the controls (standard mixture and liver pool) will be included multiple times in the randomization scheme such that sample preparation and analytical variability are constantly monitored. Furthermore, analysis of each clinical sample will be followed by at least two blank runs to prevent any carryover of metabolites between samples. The bacterial genomic DNA from feces will be extracted using MO BIO PowerSoil DNA Isolation Kit (MO BIO Laboratories). DNA extraction and 16S rRNA gene sequencing will be performed with methods consistent with those developed for the NIH-Human Microbiome Project. Briefly, the microbiome will be measured by deep sequencing of 16S rRNA genes on the Illumina MiSeq platform. 16S rRNA genes contained in every sample will be isolated by amplifying multiple regions of the 16S rRNA genes with barcoded, degenerate primers that target the V4 hypervariable domain of the gene. These primers also contain adapters for MiSeq sequencing so that the PCR products may be pooled and sequenced directly. Pooling will enable us to achieve a depth of sequencing of at least 5,000 reads per sample. Rarefaction and collector's curves of microbial community data will be constructed using sequence data for each sample to ensure that we are sampling the majority of the diversity present.

A purposeful approach to analyzing the stored blood and stool samples will be used. Initial measurements will be made on stool and blood samples obtained from a subset of the time points. Selection of additional time points for sample analysis will be made based on the initial findings. For example, if measurements made on samples obtained at weeks 1, 4 and 8 indicate that there is limited within-participant variability over an 8-week period, performing additional measurements using samples from weeks 2, 3, 5, 6, and 7 will have low priority. However, if within-participant variability is evident using the samples from weeks 1, 4 and 8, performing measurements on the weekly samples, and/or the within-week samples will be of greater interest.

# 6 Study Agent

### 6.1 Description

p-Inulin (oligofructose-enriched inulin) is a prebiotic. p-Inulin will be provided in individual packets that each contain 2 g of product. This study will utilize Prebiotin Prebiotic Fiber Stick Pac 2 g distributed by Jackson GI Medical.

#### 6.2 Treatment Regimen

All participants will take a p-inulin dose of 8 g two times per day for a total daily dose of 16 g. For each dose, the contents of four packets will be added by the participant to 100-200 ml of any type of liquid and taken orally. Treatment duration is 12 weeks. If a dose reduction of the study agent is required during the treatment phase, the investigator will instruct the participant to use only 2 packets (4 g) twice daily for a total daily dose of 8 g per day. The study agent will be discontinued if further dose reduction is required.

### 6.3 Administration of Study Agent

Study agent will be prepared by the University of Pennsylvania Investigational Drug Service (IDS), the Central Pharmacy for this study. Each study agent kit will contain a 4-week supply. The participant will receive a 4-week supply of study agent at the Week 8, 12, and 16 visits.

### 6.4 Receiving, Storing, Dispensing and Returning Study Agent

## 6.4.1 Receiving Study Product (p-Inulin) Supplies

The Central Pharmacy will distribute study agent kits to the research pharmacy at each Clinical Center. Each Clinical Center research pharmacy will be responsible for maintaining detailed records regarding the receipt of study agent. General study product accountability, participant-specific study product Accountability, and if necessary, Shipment Tracking Accountability Logs will be maintained by the site pharmacist to document study agent use. Documentation includes study product receipt, storage, dispensing, and final disposition.

### 6.4.2 Storage

The boxes containing p-inulin will be stored in a locked cabinet at the University of Pennsylvania Investigational Drug Service until shipment to the Clinical Center research pharmacy. After receipt by the Clinical Center, the study agent will be stored at the research pharmacy until distribution to the participant.

The study agent will be stored at 25°C (77°F) with excursions of 15-30°C (59-86°F) permitted.

## 6.4.3 Dispensing Study Agent

Upon enrollment of a participant, study personnel will request from the Central Pharmacy that three study agent kits are sent to the Clinical Center research pharmacy. The study agent will be dispensed by the Clinical Center research pharmacy in 4-week supplies at the Week 8, 12, and 16 visits to either an appropriate member of the research team or to the participant in accordance with Clinical Center policies and preferences.

### 6.4.4 Return or Destruction of Study Agent

Participants will return any unused study agent at the Week 12, 16, and 20 visits.

Returned product will be counted and recorded by study staff and documented on the Study Agent Dispensing and Accountability log.

At the completion of the study, there will be a final reconciliation of study agent shipped, study agent consumed, and study agent remaining. This reconciliation will be logged on the study agent reconciliation form, signed and dated. Any discrepancies noted will be investigated, resolved, and documented before the return or destruction of unused study agent. Study agent destroyed on site will be documented in the study files.

#### 6.5 Participant Adherence Monitoring

Adherence to the study agent will be assessed by counts of returned packets at the Week 12, 16, and 20 visits and from participant self-report.

### 6.6 Concomitant Therapy

Medication use (both oral and intravenous) will be collected at baseline and throughout the course of the study. Information about over the counter medications, vitamins, herbal supplements, and prebiotic and probiotic supplements in any form will also be collected. Appropriate sources for obtaining this information include the participant, the medical record, and treating clinicians.

Participants will be told not to eat probiotic yogurt throughout study participation. Participants will continue their medications including anti-hypertensive agents, phosphate binders, vitamin D preparations, erythropoietin stimulating agents, and oral or intravenous iron as prescribed by the treating physician.

Patients with chronic antibiotic use for any specified indication will not be enrolled.

### 7 Statistical Plan

## 7.1 Sample Size Determination

The target sample size is 10 participants who complete phase 1 and phase 2 and provide sufficient number of stool samples. "Sufficient" number of stool samples is defined as 2 samples during Weeks 1-4, 2 samples during Weeks 5-8, 3 samples during Weeks 9-14, and 3 samples during Weeks 15-20. Additional participants will be enrolled (up to 10 additional participants) as needed to obtain a total of 10 participants who meet the follow-up duration and sample sufficiency criteria. Participants who do not meet the sample sufficiency criteria will continue in the study and will continue to be encouraged to provide samples in accordance with the protocol schedule. Because of the high prevalence of diabetes mellitus among patients with ESRD and potential differences in the gut microbiome between patients with and without diabetes, the study will aim to have approximately 50% of participants with diabetes and 50% of participants without diabetes. Participants will be enrolled from 4 centers.

This repeated measures study design will provide important preliminary data on week-to-week variability of gut microbiome and on the effects of p-inulin on microbiome composition. Referring to relevant simulations, <sup>82</sup> the power for detecting various changes in microbiome composition based on 10 participants, before and after p-inulin treatment, can be estimated. **Figure 2** shows the power for detecting changes in community membership, evenness, richness and lineages for various effect sizes based on distance-based MANOVA analysis using different distances based on a 2D circle simulation. **Figure 3** shows the power of change of taxa clusters of various abundances based on simulating data on a phylogenetic tree. For a sample size of 10, we have adequate power to detect moderate to large effect sizes.

Based on a paired t-test, a sample size of 10 can detect an effect size smaller than 1.7 of p-inulin on metabolite changes assuming that 25 metabolites will be tested and that adjustment for multiple

comparisons will be conducted within the framework outlined by Benjamini and Hochberg for controlling the false discovery rate (FDR).<sup>83</sup> The multicenter nature of the study will provide information about the feasibility of stool sample collection for future multicenter studies of the gut microbiome.



**Figure 2. Power to Detect Composition Changes** 



Figure 3. Power to Detect Changes of Taxa Clusters

## 7.2 Missing Data

In general, missing data will not be imputed. Every effort will be made to use statistical methods that are robust to missingness, and the number of participants included with each analysis will be given with the results.

## 7.3 Statistical Methods

### 7.3.1 Sequence Data Processing

Longitudinal stool samples will be analyzed by sequencing of 16S rRNA gene tags to characterize bacterial populations. Sequence data will be processed using QIIME, augmented by the R package QIIMER (http://cran.r-project.org/web/packages/qiimer). Taxonomy will be assigned to the sequences using Ribosomal Database Project (RDP) for 16S, augmented by analysis of specific sequences using BLAST. The 16S tag sequences will be collected into operational taxonomic units (OTUs) with 97% sequence identity and samples summarized as vectors of proportions.

### 7.3.2 Analysis of Microbial Composition

Stool samples will be compared longitudinally within individual subjects, and between groups. Variability of gut microbiomes across the first 8 weeks, and during the p-inulin treatment period will be assessed at both the microbial diversity level, and the individual taxon level. The analysis will be performed at the overall microbiome composition level by calculating the alpha and beta diversities using UniFrac distances. Principal coordinate analysis (PCA) based on the UniFrac distances will be performed and used to display the samples in PCA space.

For each individual, the alpha-diversity of bacterial genera will be calculated at each time point. Alphadiversity is used to describe the structure of the bacterial community based on the number of species, and the proportion in which each species is represented in the community. The alpha diversity as a measurement will be analyzed using the repeated measurement ANOVA. To measure inter-individual variability, the beta diversity will be calculated to measure the compositional dissimilarity between two individuals at a given time point. To account for the phylogenetic tree information of the bacterial taxa, UniFrac distances (both weighted and unweighted) will be used as the beta diversity measure. Withinindividual distances and between-individual distances will be compared and clustering analysis of all the samples will be performed using the UniFrac distances. A repeated measure distance-based MANOVA will be used to assess the changes of the overall microbial compositions over time. The intraclass correlation coefficient will be determined using mixed models, with the individual as the cluster and multiple diversity observations as groups. The beta diversity will be applied with PREMANOVA and kernel-based regression in order to test the overall microbiome compositional differences between groups and over times. The genus-level analysis will be analyzed using rank-based tests using false discovery rate (FDR) control procedures for multiple comparisons to identify the bacterial genera that change their abundances over time and show different profiles between treatment/control periods. Linear mixed-effect models will also be explored after appropriate transformation of the proportional data (e.g., logistic transformation). In addition to evaluating the intra-individual and interindividual variability at the overall microbial compositional level, such variability will be evaluated at the taxon level, e.g., at each genus level. From 16S data, estimates will be obtained of the relative proportion of each of the bacterial genera observed in the data. For each bacterial taxon, a zero enriched beta regression model will be fit with random effects to assess the intra-individual and interindividual variability, both in terms of presence/absence and also the relative abundances.

The effects of p-inulin on gut microbiome compositions will be assessed using repeated measurements ANOVA with alpha-diversity as the outcome. This assesses whether p-inulin has any effect on the overall gut microbial diversity. The distance-based MANOVA will be applied to test the effect of p-inulin on overall microbial compositions, where UniFrac distances will be used. To identify the bacterial taxa that show differential abundances before and after p-inulin treatment, a zero-enriched beta regression model will be fit with random effects to take into account week-to-week variability. Similar analyses will be performed to compare the microbiome compositions between week 1 and study completion and between treatment stop and the end of study.

We will also explore various functional data analysis methods to identify the bacterial taxa with differential abundances after the p-inulin treatment, where the taxonomic profile of each individual measured over 8 weeks of time is treated as functional data. The paired functional data can be modeled with mixed effects models using basis functions or penalized splines<sup>84</sup>. We can then test the overall mean function differences before and after p-inulin treatment using a likelihood ratio test. We will consider different transformation of the proportional data before fitting the mixed effects model.

Microbiome differences between diabetic and non-diabetic participants before p-inulin treatment will be explored taking into account week-to-week variability using a mixed-effects model for alpha diversity, and a zero-enriched regression analysis for each of the taxa.

### 7.3.3 Analysis of metabolomic profile and targeted metabolites

For each of the metabolites, standard mixed-effects models will be applied to assess the intra- and interindividual variability. Nonlinear random effects models will be fit to account for possible heterogeneity in the intra-individual variance structure. Standard repeated measurement ANOVA and mixed-effect models will be applied to study change of metabolites before and after p-inulin treatment and to identify the metabolites that change after p-inulin treatment. Adjustment for multiple comparisons will be conducted within the framework outlined by Benjamini and Hochberg for controlling the false discovery rate (FDR).<sup>83</sup>

## 7.3.4 Association between microbiome composition and metabolites

Associations between microbiome and metabolites will be explored through correlation analysis and clustering analysis, focusing on the metabolites and microbial taxa that change over the study periods. Repeated measurement regression analysis of metabolite with time-varying covariates (microbiome diversity or microbial genera) will be used to identify the microbial genera that are associated with changes of metabolites due to p-inulin treatment.

#### 7.3.5 Analysis of Safety

Standard descriptive statistics will be used to summarize adverse events during the three phases (pretreatment, p-inulin treatment, and post-treatment) and graphical methods including stem-and-leaf diagrams will be used to examine distributions of adverse events. Frequencies will be compared between the treatment and non-treatment phases for the total number of events, number of participants experiencing events, events within body system categories (e.g., gastrointestinal system events), and events within severity categories.

# 8 Safety and Adverse Events

## 8.1 Definitions

Definitions are per the January 2007 Guidance on Reviewing and Reporting Unanticipated Problems Involving Risks to Participants or Others and Adverse Events, Office on Human Research Protection (OHRP) Guidance. http://www.hhs.gov/ohrp/policy/advevntguid.html

#### 8.1.1 Adverse Event

An *adverse event (AE)* is any untoward or unfavorable medical occurrence in a human study participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's involvement in the research, whether or not considered related to the participant's participation in the research.

### 8.1.2 Serious Adverse Event

A serious adverse event (SAE) is any AE that is:

- fatal or results in death
- life-threatening
- requires or prolongs hospital stay
- results in persistent or significant disability or incapacity
- results in congenital anomalies or birth defects
- an important medical event\*

#### 8.1.3 Unanticipated Problems Involving Risk to Participants or Others

An Unanticipated Problem is any incident, experience, or outcome that meets <u>all</u> of the following criteria:

- it is unexpected (in terms of nature, severity, or frequency) given the research procedures that are described in the IRB-approved research protocol and informed consent document and the characteristics of the participant population being studied;
- it is related or possibly related to participation in the research; possibly related means that there is a reasonable possibility that the incident, experience or outcome may have been caused by the procedures involved in the research, and
- it suggests that the research places participants or others at a greater risk of harm (including physical, psychological, economic, or social harm) related to the research than was previously known or recognized.

### 8.1.4 Pre-Existing Condition

A preexisting condition is one that is present at the start of the study. A preexisting condition will be recorded as an adverse event if the frequency, intensity, or the character of the condition worsens during the study period.

### 8.2 Adverse Event Reporting Period

The study period during which adverse events must be tracked and reported is defined as the period from the initiation of study procedures to study completion.

<sup>\*</sup>Important medical events are those that may not be immediately life threatening, but are clearly of major clinical significance.

### 8.2.1 Post-study Adverse Event

All unresolved adverse events will be followed by the investigator until the events are resolved, the participant is lost to follow-up, or the adverse event is otherwise explained. At the last scheduled visit, the investigator will instruct each participant to report any subsequent event(s) that the participant, or the participant's personal physician, believes might reasonably be related to participation in this study. The investigator will notify the Data Coordinating Center (DCC) of any death or adverse event occurring at any time after a participant has discontinued or terminated study participation that may reasonably be related to the study.

### 8.3 Recording of Adverse Events

At each contact with the participant, the investigator or site designee will seek information on adverse events by specific questioning and, as appropriate, by examination. Information on adverse events will be recorded in the source document, and also on the adverse event log case report form (CRF). All signs, symptoms, and abnormal diagnostic procedure results relating to the same event will be recorded under one diagnosis name.

#### 8.3.1 Anticipated Adverse Events

The following adverse events are anticipated in the hemodialysis population and are not considered Unanticipated Problems. Note that the designation as "Anticipated" does not imply that the event is not an SAE but relates to the regulatory definition of Unanticipated Problems as provided in Section 8.1.3.

- Death
- Coronary Ischemia including:
  - o Unstable angina
  - Acute MI
  - Coronary revascularization
- Heart failure hospitalization or exacerbation
- Cardiac arrest
- Cardiac arrhythmia (ventricular or atrial)
- Peripheral vascular revascularization
- Amputation
- Hypotension
- Vomiting
- Vascular Access Events Including:
  - Catheter exchange, removal or declotting
  - Arteriovenous graft or fistula complications
    - Clotting
    - Stenosis
    - Revascularization
    - Infection
- Infections Including:
  - Pneumonia

#### Bacteremia

## Hemodialysis vascular access infection Non-Reportable Events

The hemodialysis population is characterized by frequent laboratory testing and a high rate of peridialytic hypotensive events requiring change in the dialysis prescription, adjustment of dry weight or change in dialysis-related medications. Due to the unique nature of this population, the following events are considered routine aspects of chronic dialysis therapy and they will not be considered to meet the criteria of SAE in this study except as noted:

- Anemia—will be reported only when hemoglobin <8.0 mg/dL</li>
- Hyperphosphatemia-will be reported only when phosphorus >9.5 mg/dL
- Hypocalcemia-will be reported only when serum calcium < 7.0 mg/dL</li>
- Hypercalcemia-will be reported only when serum calcium >11.0 mg/dL
- Hyperparathyroidism-will be reported only when PTH>1000 pg/mL
- Hypotension-will be reported only when requiring emergency room visit or hospitalization

## 8.4 Reporting of Serious Adverse Events and Unanticipated Problems

Study sites are required to report SAEs to the DCC within 24 hours of first knowledge of the event. To report such events, an SAE form will be completed by the investigator and faxed or emailed to the DCC. The DCC will facilitate the timely medical review and reporting of the event and updates to the NIDDK and the Data and Safety Monitoring Board (DSMB) in accordance with DSMB-approved study policies and regulatory requirements (see Section 8.5.1 for details of the DSMB).

The investigator will keep a copy of the SAE form on file at the study site. At the time of the initial report, the following information should be provided:

- Study identifier
- Study Center
- Participant number
- A description of the event
- Date of onset
- Current status

- Whether study treatment was discontinued
- The reason why the event is classified as serious
- Investigator assessment of the association between the event and study participation

Within the following 7 days, the investigator will provide further information on the SAE or the unanticipated problem in the form of a written narrative. This should include a copy of the completed SAE form, and any other diagnostic information that will assist the understanding of the event. Significant new information on ongoing serious adverse events should be provided promptly to the DCC.

If a participant becomes pregnant while participating in the study it will be reported as an adverse event and will trigger the collection of additional documentation about the pregnancy. Pregnancy outcomes will be collected, including the outcome of the infant and if the pregnancy was terminated. This information will be submitted to the University of Pennsylvania IRB, and to the local site IRB as required.

SAEs that are still ongoing at the end of the study period must be followed up to determine the final outcome. Any SAE that occurs after the study period and is considered to be possibly related to the study treatment or study participation should be recorded and reported immediately.

### 8.4.1 Investigator Reporting to the IRB

Site investigators will report SAEs and Unanticipated problems to their IRB in accordance with the reporting requirements of the local IRB or with the Office of Human Research Protections (OHRP) guidelines, whichever is sooner. OHRP recommends that:

- 1) Unanticipated problems that are serious adverse events should be reported to the IRB within 1 week of the investigator becoming aware of the event; and
- 2) Any other unanticipated problem should be reported to the IRB within 2 weeks of the investigator becoming aware of the problem.

### **Reporting Process**

Unanticipated problems posing risks to participants or others as noted above will be reported using the appropriate IRB-designated form or as a written report of the event (including a description of the event with information regarding its fulfillment of the above criteria, follow-up/resolution and need for revision to consent form and/or other study documentation).

Copies of each report and documentation of IRB notification and receipt will be maintained in the Clinical Center Investigator's study file.

#### **Other Reportable Events:**

- Any adverse event that would cause the sponsor to modify the protocol or informed consent form, or would prompt other action by the IRB to assure protection of human participants.
- Information that indicates a change to the risks or potential benefits of the research, in terms of severity or frequency.
- Breach of confidentiality
- Change to the protocol made without prior IRB review to eliminate apparent immediate hazard to a research participant.
- Incarceration of a participant when the research was not previously approved under Subpart C
  and the investigator believes it is in the best interest of the participant to remain in the study.
- Complaint of a participant when the complaint indicates unexpected risks or the complaint cannot be resolved by the research team.
- Protocol violation (meaning an accidental or unintentional deviation from the IRB approved protocol) that in the opinion of the investigator placed one or more participants at increased risk, or affects the rights or welfare of participants.

#### 8.4.2 DCC Notification to Participating Investigators

The DCC will notify all Clinical Center principal investigators, in a written safety report, of any adverse event that meets the criteria of an unanticipated and related event as described in **Section 8.1.3**.

### 8.5 Medical Monitoring

Each Clinical Center Principal Investigator will be responsible for overseeing the safety of the study at his/her site. This safety monitoring will include careful assessment and appropriate reporting of adverse events as noted above, as well as the construction and implementation of a site data and safety-monitoring plan. Medical monitoring will include a regular assessment of the number and type of serious adverse events.

### 8.5.1 Independent Data and Safety Monitoring Board (DSMB)

The information provided in this section of the protocol is a general description of the DSMB responsibilities and processes. A DSMB charter for the Hemodialysis Novel Therapies Consortium includes additional detail. The NIDDK DSMB charter is provided as an attachment in **Section 15**.

A DSMB has been established by the NIDDK and provides input to the Institute. The DSMB is comprised of individuals with expertise in clinical trials design and methodology, biostatistics, clinical nephrology and other relevant medical specialties. The DSMB members are not affiliated with the study and are appointed by the NIDDK. DSMB members will be free of conflicts of interest that could be affected by the outcomes of the study. During the study, DSMB members who develop real or perceived conflicts of interest that impact objectivity will disclose them to NIDDK project officers, who will arrange for replacement of the member, if indicated.

The DSMB will review the protocol before initiation of the study. After initial approval during the course of the study, the primary responsibilities of the DSMB will be to:

- Review safety data and provide input to protect the safety of the study participants;
- Provide input on major changes to the research protocol and plans for data and safety monitoring;
- Provide input on the progress of the study, including periodic assessments of data quality and timeliness, participant recruitment, accrual and retention, participant risk versus benefit, performance of the study sites, and other factors that may affect study outcomes;
- Consider factors external to the study when relevant information becomes available, such as scientific or therapeutic developments that may have an impact on the need for continuation of the study, safety of the participants or the ethics of the study;
- Provide input on modification of the study protocol or possible early termination of the study because of attainment of study objectives, safety concerns, or inadequate performance (such as enrollment and retention problems).

## 9 Data management

An internet-based registration system designed by the DCC will be used for all of the pilot and feasibility studies of the Hemodialysis Novel Therapies Consortium in order to promote uniformity across studies. The central registration system will include a randomization module for each study that will confirm eligibility. Central participant registration will also allow the DCC to generate recruitment reports across concurrent studies.

An Oracle Clinical data management system (DMS) designed by the DCC will be used for the collection, storage and management of data. Site personnel will enter data directly using Oracle Clinical Remote Data Capture. Electronic case report forms (eCRFs) will incorporate range and logical edit checks, both within and across forms. Data entry will be followed daily with manual and programmed checks and edits for errors and omissions.

### 9.1 Data Quality

The DCC will collaborate with the Clinical Center investigators to establish parameters for primary and secondary outcomes, safety, and descriptive values. The data management team will use a data validation plan, rule set specifications, and programming logic to implement data validation rules. The DCC staff will interact with Clinical Center study staff to verify queried data and track all queries to resolution.

### 9.1.1 Quality Control Activities

The Quality Control Committee and the DCC will develop a quality assurance and control plan that ensures that study data are as precise and reliable as possible.

<u>Manual of Procedures</u> (MOP) – The MOP will describe the sequence of study conduct and provide detailed instruction for the performance of screening, baseline, enrollment, treatment allocation and follow-up procedures. The MOP will provide instruction in case report form (CRF) completion, use of the electronic DMS, and collection, documentation and transfer of specimens and tests to central laboratories.

<u>Training and certification procedures</u> – The DCC will conduct a training session before the study starts to train and certify personnel in the performance of study procedures.

<u>Site visits</u> – Site visits will be conducted as outlined in the Study Monitoring Plan. Findings from site visits will be used to resolve problems and develop corrective action plans.

External data sources – The DCC will monitor quality control of data received from central laboratories.

<u>Internal quality control procedures</u> – A data validation plan, rule set specifications, and programming logic to implement data validation rules will be implemented.

#### 9.1.2 Routine reports

The DCC will develop a set of standard enrollment, tracking, quality review, and safety monitoring reports. Adverse event reports, DSMB reports and reports for statistical analysis will be developed and produced on an appropriate schedule.

#### 9.2 Data Security

The DMS will be designed to prevent unauthorized access to study data and to prevent data loss due to equipment failure or catastrophic events. The procedures to do so encompass user account management, user privilege assignment, data loss prevention (database backup), and DMS change management. User access will be controlled by assignment of confidential usernames and passwords.

Study data collected at the Clinical Centers will be entered into Oracle Clinical. This DMS uses a secure connection between the client browser at the Clinical Center and the web server at the DCC. Data transmitted over this connection is authenticated by the use of digital certificates and is encrypted as it travels the Internet to the DCC.

Where applicable, electronic files containing data from hand held devices and central laboratories will be transferred to the DCC using secure File Transfer Protocol (FTP) technology. The DCC team will maintain a secure FTP server. The files transmitted using this method will be encrypted during the exchange.

### 9.2.1 Confidentiality

Information about study participants will be kept confidential and managed according to the requirements of the Health Insurance Portability and Accountability Act of 1996 (HIPAA). Those regulations require a signed participant authorization informing the participant of the following:

- What protected health information (PHI) will be collected from participants in this study
- Who will have access to that information and why
- Who will use or disclose that information
- The rights of a research participant to revoke their authorization for use of their PHI.

In the event that a participant revokes authorization to collect or use PHI, the investigator, by regulation, retains the ability to use all information collected before the revocation of participant authorization. For participants that have revoked authorization to collect or use PHI, attempts should be made to obtain permission to collect at least vital status (i.e. that the participant is alive) at the end of their scheduled study period.

### 9.3 Source Documents

Source data is all information, original records of clinical findings, observations, or other activities in a research study necessary for the reconstruction and evaluation of the study. Source data are contained in source documents. Examples of these original documents, and data records include: dialysis unit records, hospital records, clinical and office charts, laboratory reports, memoranda, participant diaries or evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, copies or transcriptions certified after verification as being accurate and complete, microfiches, photographic negatives, microfilm or magnetic media, x-rays, participant files, and records kept at the pharmacy, at the laboratories, and at medico-technical departments involved in the clinical trial.

## 9.3.1 Case Report Forms

The study CRF is the primary data collection instrument for the study. All data requested on the CRF will be recorded. All missing data will be explained. "N/D" will be used to indicate on the CRF that a procedure was not done or a question was not asked rather than leaving a space blank. "N/A" will be used to indicate that an item is not applicable to the individual case. All entries will be printed legibly in black ink. If any entry error has been made, to correct such an error, a single straight line will be drawn through the incorrect entry and the correct data will be entered above it. All such changes will be

initialed and dated. Erasing or white-out will not be used for errors. For clarification of illegible or uncertain entries, the clarification will be printed above the item, and the clarification will be initialed and dated.

### 9.3.2 Maintaining Anonymity of Submitted Medical Records

Clinical site personnel will de-identify all medical records before sending them to the DCC by removing any PHI. Upon receipt, DCC personnel will review the records to ensure that no PHI is visible.

### 9.3.3 Data Sharing

Research results will be made available to the scientific community and public in a timely manner. The primary method by which data will be shared with the scientific community will be through peer-reviewed publications and presentation at scientific and professional society meetings. In addition, data and results will be submitted to the NIH in the annual progress reports required under the terms and conditions of the funding award. This study will also be registered with clinicaltrials gov before initiation.

Data from the study will be submitted to the NIDDK Data Repository in accordance with the NIDDK Data Sharing policy. The policy requires that data sets be transferred no later than 2 years after study completion or 1 year after publication of the primary results, whichever comes first. Through the repository, the study data will be made available to external investigators.

#### 9.3.4 Records Retention

The site investigators will retain study documents, including participant files and Regulatory Binders, for at least 5 years after the close of the study, or longer depending on site institutional requirements.

# 10 Study Monitoring, Auditing, and Inspecting

## 10.1 Study Monitoring Plan

A monitoring plan that may include formal visits to the Clinical Centers by members of the Consortium (DCC, Clinical Center investigators and study coordinators, and NIDDK representatives) will be developed by the Consortium Executive Committee. Clinical Center investigators will allocate adequate time for such monitoring activities. The Principal Investigator will also ensure that the monitor and other compliance or quality assurance reviewers are given access to study-related documents and study-related facilities (e.g. pharmacy, diagnostic laboratory, etc.), and have adequate space to conduct the monitoring visit.

### 10.2 Auditing and Inspecting

The DCC and Clinical Center investigators will permit study-related monitoring, audits, and inspections by the IRB, the NIH, government regulatory bodies, and University compliance and quality assurance groups of all study related documents (e.g. source documents, regulatory documents, data collection instruments, study data etc.). The DCC and Clinical Center investigators will ensure the capability for inspections of applicable study-related facilities (e.g. pharmacy, diagnostic laboratory, etc.).

Participation as an investigator in this study implies acceptance of potential inspection by government regulatory authorities and applicable institution compliance and quality assurance offices.

# 11 Ethical Considerations

This study will be conducted according to US and international standards of Good Clinical Practice, all applicable government regulations and research policies and procedures in effect at the Institutions where this study is implemented.

This protocol and any amendments will be submitted to a properly constituted independent IRB, in agreement with local legal prescriptions, for formal approval of the study. The decision of the IRB concerning the conduct of the study will be made in writing to the Clinical Center investigator and a copy of this decision will be provided to the DCC before commencement of the study at the site.

All study participants will be provided a consent form describing the study and providing sufficient information to make an informed decision about participating in the study. The consent form will be submitted with the protocol for review and approval by the IRB. The formal consent of a participant, using the IRB-approved consent form, must be obtained before that participant undergoes any study procedure. The consent form must be signed by the participant or legally acceptable surrogate, and the investigator-designated research professional obtaining the consent.

# 12 Study Finances

### 12.1 Funding Source

This study is financed through grants from the National Institute of Diabetes and Digestive and Kidney Diseases of the U.S. National Institutes of Health.

#### 12.2 Conflict of Interest

All investigators will follow the conflict of interest policies of the National Institutes of Health as well as their home institution. Any investigator who has a potential conflict of interest with this study (patent ownership, royalties, or financial gain greater than the minimum allowable by their institution, etc.) must have the conflict reviewed by a properly constituted Conflict of Interest Committee with a Committee-sanctioned conflict management plan that has been reviewed and approved by the study sponsor before participation in this study.

#### 12.3 Participant Stipends or Payments

Participants will be compensated for participating in the study. Compensation approaches will be determined by the Clinical Centers and approved by the local IRB.

## 13 Publication Plan

Neither the complete, nor any part of, the results of the study carried out under this protocol, nor any of the information provided by the Hemodialysis Novel Therapies Consortium for the purposes of performing the study, will be published or passed on to any third party without the consent of the

Consortium Executive Committee and Steering Committee. Any investigator involved with this study is obligated to provide the DCC with results of all study-related testing and all data derived from the study.

## 14 References

- 1. Kimmel PL, Phillips TM, Simmens SJ, et al. Immunologic function and survival in hemodialysis patients. *Kidney Int* 1998;54(1):236-244.
- 2. Zimmermann J, Herrlinger S, Pruy A, Metzger T, Wanner C. Inflammation enhances cardiovascular risk and mortality in hemodialysis patients. *Kidney Int* 1999;55(2):648-658.
- 3. Ioannidou E, Swede H, Dongari-Bagtzoglou A. Periodontitis predicts elevated C-reactive protein levels in chronic kidney disease. *J Dent Res* 2011;90(12):1411-1415.
- 4. Goncalves S, Pecoits-Filho R, Perreto S, et al. Associations between renal function, volume status and endotoxaemia in chronic kidney disease patients. *Nephrol Dial Transplant* 2006;21(10):2788-2794.
- 5. Ramos LF, Shintani A, Ikizler TA, Himmelfarb J. Oxidative stress and inflammation are associated with adiposity in moderate to severe CKD. *J Am Soc Nephrol* 2008;19(3):593-599.
- 6. Safieh-Garabedian B, Poole S, Haddad JJ, Massaad CA, Jabbur SJ, Saade NE. The role of the sympathetic efferents in endotoxin-induced localized inflammatory hyperalgesia and cytokine upregulation. *Neuropharmacology* 2002;42(6):864-872.
- 7. Sterling KA, Eftekhari P, Girndt M, Kimmel PL, Raj DS. The immunoregulatory function of vitamin D: implications in chronic kidney disease. *Nat Rev Nephrol* 2012;8(7):403-412.
- 8. Vaziri ND. CKD impairs barrier function and alters microbial flora of the intestine: a major link to inflammation and uremic toxicity. *Curr Opin Nephrol Hypertens* 2012;21(6):587-592.
- 9. Vaziri ND, Wong J, Pahl M, et al. Chronic kidney disease alters intestinal microbial flora. *Kidney Int* 2013;83(2):308-315.
- 10. Raj DS, Carrero JJ, Shah VO, et al. Soluble CD14 levels, interleukin 6, and mortality among prevalent hemodialysis patients. *Am Journal Kidney Dis* 2009;54(6):1072-1080.
- 11. Raj DS, Shah VO, Rambod M, Kovesdy CP, Kalantar-Zadeh K. Association of soluble endotoxin receptor CD14 and mortality among patients undergoing hemodialysis. *Am J Kidney Dis* 2009;54(6):1062-1071.
- 12. Ramezani A, Raj DS. The gut microbiome, kidney disease, and targeted interventions. *J Am Soc Nephrol* 2014;25(4):657-670.
- 13. Backhed F, Ding H, Wang T, et al. The gut microbiota as an environmental factor that regulates fat storage. *Proc Natl Acad Sci USA* 2004;101(44):15718-15723.
- 14. Tang WH, Wang Z, Levison BS, et al. Intestinal microbial metabolism of phosphatidylcholine and cardiovascular risk. *N Engl J Med* 2013;368(17):1575-1584.
- 15. Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. *Nature* 2006;444(7122):1027-1031.
- 16. Hooper LV, Midtvedt T, Gordon JI. How host-microbial interactions shape the nutrient environment of the mammalian intestine. *Annu Rev Nutr* 2002;22:283-307.
- 17. Hill MJ. Intestinal flora and endogenous vitamin synthesis. *Eur J Cancer Prev* 1997;6 Suppl 1:S43-45.
- 18. Hylemon PB, Harder J. Biotransformation of monoterpenes, bile acids, and other isoprenoids in anaerobic ecosystems. *FEMS Microbiol Rev* 1998;22(5):475-488.
- 19. Duncan SH, Richardson AJ, Kaul P, Holmes RP, Allison MJ, Stewart CS. Oxalobacter formigenes and its potential role in human health. *App Environmen Microbiol* 2002;68(8):3841-3847.
- 20. Braun-Fahrlander C, Riedler J, Herz U, et al. Environmental exposure to endotoxin and its relation to asthma in school-age children. *N Engl J Med* 2002;347(12):869-877.
- 21. Simenhoff ML, Dunn SR, Zollner GP, et al. Biomodulation of the toxic and nutritional effects of small bowel bacterial overgrowth in end-stage kidney disease using freeze-dried Lactobacillus acidophilus. *Miner Electrolyte Metab* 1996;22(1-3):92-96.
- 22. Hida M, Aiba Y, Sawamura S, Suzuki N, Satoh T, Koga Y. Inhibition of the accumulation of uremic toxins in the blood and their precursors in the feces after oral administration of Lebenin, a lactic acid bacteria preparation, to uremic patients undergoing hemodialysis. *Nephron.* 1996;74(2):349-355.
- 23. Kang JY. The gastrointestinal tract in uremia. Dig Dis Sci 1993;38(2):257-268.
- 24. Vaziri ND, Dure-Smith B, Miller R, Mirahmadi MK. Pathology of gastrointestinal tract in chronic hemodialysis patients: an autopsy study of 78 cases. *AmJ Gastroenterol* 1985;80(8):608-611.

- 25. Kalantar-Zadeh K, Kopple JD, Deepak S, Block D, Block G. Food intake characteristics of hemodialysis patients as obtained by food frequency questionnaire. *J Ren Nutr* 2002;12(1):17-31.
- 26. Hatch M, Freel RW, Vaziri ND. Intestinal excretion of oxalate in chronic renal failure. *J Am Soc Nephrol* 1994;5(6):1339-1343.
- 27. Schena FP. Management of patients with chronic kidney disease. *Intern Emerg Med* 2011;6 Suppl 1:77-83.
- 28. Jakobsson HE, Jernberg C, Andersson AF, Sjolund-Karlsson M, Jansson JK, Engstrand L. Short-term antibiotic treatment has differing long-term impacts on the human throat and gut microbiome. *PloS One* 2010;5(3):e9836.
- 29. Jernberg C, Lofmark S, Edlund C, Jansson JK. Long-term impacts of antibiotic exposure on the human intestinal microbiota. *Microbiology* 2010;156(Pt 11):3216-3223.
- 30. Lefebvre HP, Ferre JP, Watson AD, et al. Small bowel motility and colonic transit are altered in dogs with moderate renal failure. *Am J Physiol. Regul Integr Comp Physiol* 2001;281(1):R230-238.
- 31. Wu MJ, Chang CS, Cheng CH, et al. Colonic transit time in long-term dialysis patients. *Am J Kidney Dis* 2004;44(2):322-327.
- 32. Goraya N, Wesson DE. Dietary management of chronic kidney disease: protein restriction and beyond. *Curr Opin Nephrol Hypertens* 2012;21(6):635-640.
- 33. Goraya N, Wesson DE. Acid-base status and progression of chronic kidney disease. *Curr Opin Nephrol Hypertens* 2012;21(5):552-556.
- 34. Kooman JP, van der Sande FM, Leunissen KM. Role of sodium and volume in the pathogenesis of hypertension in dialysis patients. Reflections on pathophysiological mechanisms. *Blood Purif* 2004;22(1):55-59.
- 35. Sato Y, Takatsu Y, Kataoka K, et al. Serial circulating concentrations of C-reactive protein, interleukin (IL)-4, and IL-6 in patients with acute left heart decompensation. *Clin Cardiol* 1999;22(12):811-813.
- 36. Niebauer J, Volk HD, Kemp M, et al. Endotoxin and immune activation in chronic heart failure: a prospective cohort study. *Lancet* 1999;353(9167):1838-1842.
- 37. Werner T, Wagner SJ, Martinez I, et al. Depletion of luminal iron alters the gut microbiota and prevents Crohn's disease-like ileitis. *Gut* 2011;60(3):325-333.
- 38. Liguori L. Iron protein succinylate in the treatment of iron deficiency: controlled, double-blind, multicenter clinical trial on over 1,000 patients. *Int J Clin Pharmacol Ther Toxicol* 1993;31(3):103-123.
- 39. Dou L, Cerini C, Brunet P, et al. P-cresol, a uremic toxin, decreases endothelial cell response to inflammatory cytokines. *Kidney Int* 2002:62(6):1999-2009.
- 40. Cerini C, Dou L, Anfosso F, et al. P-cresol, a uremic retention solute, alters the endothelial barrier function in vitro. *Thromb Haemost* 2004;92(1):140-150.
- 41. Aronov PA, Luo FJ, Plummer NS, et al. Colonic contribution to uremic solutes. *J Amer Soc Nephrol* 2011;22(9):1769-1776.
- 42. Magnusson M, Magnusson KE, Sundqvist T, Denneberg T. Impaired intestinal barrier function measured by differently sized polyethylene glycols in patients with chronic renal failure. *Gut* 1991;32(7):754-759.
- 43. Wang F, Zhang P, Jiang H, Cheng S. Gut bacterial translocation contributes to microinflammation in experimental uremia. *Dig Dis Sci* 2012;57(11):2856-2862.
- 44. Meijers BK, Bammens B, De Moor B, Verbeke K, Vanrenterghem Y, Evenepoel P. Free p-cresol is associated with cardiovascular disease in hemodialysis patients. *Kidney Int* 2008;73(10):1174-1180.
- 45. Bammens B, Evenepoel P, Keuleers H, Verbeke K, Vanrenterghem Y. Free serum concentrations of the protein-bound retention solute p-cresol predict mortality in hemodialysis patients. *Kidney Int* 2006;69(6):1081-1087.
- 46. Stoll LL, Denning GM, Weintraub NL. Potential role of endotoxin as a proinflammatory mediator of atherosclerosis. *Arterioscl Thromb Vasc Biol* 2004;24(12):2227-2236.
- Wiedermann CJ, Kiechl S, Dunzendorfer S, et al. Association of endotoxemia with carotid atherosclerosis and cardiovascular disease: prospective results from the Bruneck Study. *J Am Coll Cardiol* 1999;34(7):1975-1981.

- 48. Pugin J, Heumann ID, Tomasz A, et al. CD14 is a pattern recognition receptor. *Immunity* 1994;1(6):509-516.
- 49. Gibson GR, Beatty ER, Wang X, Cummings JH. Selective stimulation of bifidobacteria in the human colon by oligofructose and inulin. *Gastroenterology* 1995;108(4):975-982.
- 50. Martinez I, Lattimer JM, Hubach KL, et al. Gut microbiome composition is linked to whole grain-induced immunological improvements. *ISME J* 2013;7(2):269-280.
- 51. Ewaschuk JB, Diaz H, Meddings L, et al. Secreted bioactive factors from Bifidobacterium infantis enhance epithelial cell barrier function. *Am J Physiol Gastrointest Liver Physiolphysiol* Nov 2008:295(5):G1025-1034.
- 52. Furrie E, Macfarlane S, Kennedy A, et al. Synbiotic therapy (Bifidobacterium longum/Synergy 1) initiates resolution of inflammation in patients with active ulcerative colitis: a randomised controlled pilot trial. *Gut* 2005;54(2):242-249.
- 53. Kelly D, Conway S, Aminov R. Commensal gut bacteria: mechanisms of immune modulation. *Trends Immunol* 2005;26(6):326-333.
- 54. Mazmanian SK, Liu CH, Tzianabos AO, Kasper DL. An immunomodulatory molecule of symbiotic bacteria directs maturation of the host immune system. *Cell* 2005;122(1):107-118.
- 55. Rakoff-Nahoum S, Paglino J, Eslami-Varzaneh F, Edberg S, Medzhitov R. Recognition of commensal microflora by toll-like receptors is required for intestinal homeostasis. *Cell* 2004;118(2):229-241.
- 56. Cani PD, Neyrinck AM, Fava F, et al. Selective increases of bifidobacteria in gut microflora improve high-fat-diet-induced diabetes in mice through a mechanism associated with endotoxaemia. *Diabetologia* 2007;50(11):2374-2383.
- 57. Nakabayashi I, Nakamura M, Kawakami K, et al. Effects of synbiotic treatment on serum level of p-cresol in haemodialysis patients: a preliminary study. *Nephrol Dial Transplant* 2011;26(3):1094-1098.
- 58. Meijers BK, De Preter V, Verbeke K, Vanrenterghem Y, Evenepoel P. p-Cresyl sulfate serum concentrations in haemodialysis patients are reduced by the prebiotic oligofructose-enriched inulin. *Nephrol Dial Transplant* 2010;25(1):219-224.
- 59. Roberfroid MB, Van Loo JA, Gibson GR. The bifidogenic nature of chicory inulin and its hydrolysis products. *J Nutr* 1998;128(1):11-19.
- 60. Roberfroid MB. Introducing inulin-type fructans. *Br J Nutr.* 2005;93 Suppl 1:S13-25.
- 61. Kelly G. Inulin-type prebiotics: a review. (Part 2). Altern Med Rev 2009;14(1):36-55.
- 62. Bouhnik Y, Raskine L, Simoneau G, Paineau D, Bornet F. The capacity of short-chain fructooligosaccharides to stimulate faecal bifidobacteria: a dose-response relationship study in healthy humans. *Nutr J* 2006;5:8.
- 63. Carabin IG, Flamm WG. Evaluation of safety of inulin and oligofructose as dietary fiber. *Regul Toxicol Pharmacol* 1999:30(3):268-282.
- 64. Dewulf EM, Cani PD, Claus SP, et al. Insight into the prebiotic concept: lessons from an exploratory, double blind intervention study with inulin-type fructans in obese women. *Gut* 2013;62(8):1112-1121.
- 65. Kellow NJ, Coughlan MT, Reid CM. Metabolic benefits of dietary prebiotics in human subjects: a systematic review of randomised controlled trials. *Br.J Nutr* 2013:1-15.
- 66. Gori A, Rizzardini G, Van't Land B, et al. Specific prebiotics modulate gut microbiota and immune activation in HAART-naive HIV-infected adults: results of the "COPA" pilot randomized trial. *Mucosal.lmmunol* 2011;4(5):554-563.
- 67. Monachese M, Cunningham-Rundles S, Diaz MA, et al. Probiotics and prebiotics to combat enteric infections and HIV in the developing world: a consensus report. *Gut Microbes* 2011;2(3):198-207.
- 68. Scaldaferri F, Gerardi V, Lopetuso LR, et al. Gut microbial flora, prebiotics, and probiotics in IBD: their current usage and utility. *Biomed.Res.Int* 2013;2013:435268.
- 69. Bouhnik Y, Achour L, Paineau D, Riottot M, Attar A, Bornet F. Four-week short chain fructooligosaccharides ingestion leads to increasing fecal bifidobacteria and cholesterol excretion in healthy elderly volunteers. *Nutr.J* 2007;6:42.
- 70. Garcia-Peris P, Velasco C, Lozano MA, et al. Effect of a mixture of inulin and fructo-oligosaccharide on Lactobacillus and Bifidobacterium intestinal microbiota of patients receiving radiotherapy: a randomised, double-blind, placebo-controlled trial. *Nutr Hosp* 2012;27(6):1908-1915.

- 71. Dehghan P, Gargari BP, Jafar-Abadi MA, Aliasgharzadeh A. Inulin controls inflammation and metabolic endotoxemia in women with type 2 diabetes mellitus: a randomized-controlled clinical trial. *Int.J Food Sci.Nutr* 2013; 65(1):117-123.
- 72. de Preter V, Vanhoutte T, Huys G, Swings J, Rutgeerts P, Verbeke K. Baseline microbiota activity and initial bifidobacteria counts influence responses to prebiotic dosing in healthy subjects. *Aliment Pharmacol Ther* 2008;27(6):504-513.
- 73. Schiffrin EJ, Thomas DR, Kumar VB, et al. Systemic inflammatory markers in older persons: the effect of oral nutritional supplementation with prebiotics. *J Nutr Health Aging* 2007;11(6):475-479.
- 74. Kotzampassi K, Giamarellos-Bourboulis EJ, Voudouris A, Kazamias P, Eleftheriadis E. Benefits of a synbiotic formula (Synbiotic 2000Forte) in critically III trauma patients: early results of a randomized controlled trial. *World J Surg* 2006;30(10):1848-1855.
- 75. Bouhnik Y, Raskine L, Simoneau G, et al. The capacity of nondigestible carbohydrates to stimulate fecal bifidobacteria in healthy humans: a double-blind, randomized, placebo-controlled, parallel-group, dose-response relation study. *Am J Clin Nutr* 2004;80(6):1658-1664.
- 76. Bouhnik Y, Vahedi K, Achour L, et al. Short-chain fructo-oligosaccharide administration dose-dependently increases fecal bifidobacteria in healthy humans. *J Nutr* 1999;129(1):113-116.
- 77. Meijers BK, Bammens B, De MB, Verbeke K, Vanrenterghem Y, Evenepoel P. Free p-cresol is associated with cardiovascular disease in hemodialysis patients. *Kidney Int* 2008;73(10):1174-1180.
- 78. Rao AV. Dose-response effects of inulin and oligofructose on intestinal bifidogenesis effects. *J Nutr* 1999;129(7 Suppl):1442S-1445S.
- 79. Briet F, Achour L, Flourie B, et al. Symptomatic response to varying levels of fructooligosaccharides consumed occasionally or regularly. *European J Clin Nutr* 1995;49(7):501-507.
- 80. Bruhwyler J, Carreer F, Demanet E, Jacobs H. Digestive tolerance of inulin-type fructans: a double-blind, placebo-controlled, cross-over, dose-ranging, randomized study in healthy volunteers. *Int J Food Sci Nutr* 2009;60(2):165-175.
- 81. Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. *Dig Dis Sci* 1988;33(2):129-134.
- 82. Chen J, Bittinger K, Charlson ES, et al. Associating microbiome composition with environmental covariates using generalized UniFrac distances. *Bioinformatics* 2012;28(16):2106-2113.
- 83. Benjamini Y, Hochberg Y. Controlling the false discovery rate: a practical and powerful approach to multiple testing. *J R Stat Soc Ser B-Methodol* 1995;57(1):289-300.
- 84. Zhou L, Huang J, Carrol RJ. Joine modeling of paired sparse functional data using principal components. *Biometrika* 2008:95:601-619.
- 85. Davidian M, Giltinan D. Some simple methods for estimating intra-individual variablity in nonlinear mixed effects models. *Biometrics* 1993;49:59-73

# 15 Attachments

# 15.1 Study Procedures

| | SCRE | ENING | Observation with no treatment | | | | TREATMENT PHASE WEEKS 9-20 | | | | | | | Observation with no treatment | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Pre<br>screening | Screening<br>Visit <sup>1</sup> | Baseline<br>Week 1 | Weeks<br>2-3 | Week<br>4 | Weeks<br>5-7 | Week<br>8 | Week<br>9 | Weeks<br>10-11 | Week<br>12 | Weeks<br>13-15 | Week<br>16 | Weeks<br>17-19 | Week<br>20 | Week<br>21 | Weeks<br>22-23 | Week<br>24 | Weeks<br>25-27 | Week<br>28 |
| Preliminary eligibility assessment | Х | | | | | | | | | | | | | | | | | | |
| Informed consent | | X | | | | | | | | | | | | | | | | | |
| Confirm eligibility | | Х | Х | | | | | | | | | | | | | | | | |
| Demographic info & medical history | | Х | | | | | | | | | | | | | | | | | |
| Concomitant medications | | X | Х | | Χ | | Χ | | | Χ | | Χ | | Х | | | Χ | | Х |
| Serum pregnancy | | X | | | | | | | | | | | | | | | | | |
| Blood specimen collection <sup>2</sup> | | | Х | Χ | Χ | Х | Χ | Χ | Х | Χ | Х | Χ | Χ | Χ | Х | Х | Χ | Х | Х |
| Stool sample collection | | | 3 <b>X</b> | 3 <b>X</b> | 3 <b>X</b> | 3 <b>X</b> | <sup>4</sup> X | <sup>4</sup> X | 3 <b>X</b> | 3 <b>X</b> | 3 <b>X</b> | 3 <b>X</b> | 3 <b>X</b> | <sup>4</sup> X | <sup>4</sup> X | 3 <b>X</b> | 3 <b>X</b> | 3 <b>X</b> | 3 <b>X</b> |
| Antibiotic use review (weekly) | | | Х | Χ | Χ | Х | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Х | Х | Χ | Х | Χ |
| GI symptom assessment | | | Х | | Χ | | Х | | | Х | | Χ | | Х | | | Х | | Χ |
| Food frequency questionnaire | | | Х | | | | Χ | | | | | | | Χ | | | | | Χ |
| Review adverse events | | | | | Χ | | Х | | | Х | | Χ | | Χ | | | Х | | Χ |
| Follow-up visit | | | | | Х | | Х | | | Х | | Х | | X | | | Х | | Х |
| Dispense study medication | | | | | | | Х | | | Х | | Χ | | | | | | | |
| Reconcile study medication | | | | | | | | | | Х | | Χ | | Χ | | | | | |
| Dose adjustment (prn) | | | | | | | | | 1 | | Х | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Screening and baseline activities can be performed at two separate visits or as one visit

<sup>&</sup>lt;sup>2</sup> Hemoglobin results from the dialysis unit patient record must be reviewed before each blood draw. If this result is less than 9.0 g/dl, blood will not be collected until the hemoglobin value is 9.0 g/dl or greater.

<sup>&</sup>lt;sup>3</sup> Collect 1x per week

<sup>&</sup>lt;sup>4</sup> Collect 2x per week

#### 15.2 DSMB Charter

## Data and Safety Monitoring Board (DSMB) Charter Hemodialysis Novel Therapies Consortium

The Data and Safety Monitoring Board (DSMB) will act in an advisory capacity to the National Institute of Diabetes, Digestive and Kidney Diseases (NIDDK) to monitor patient safety and evaluate the efficacy of the interventions. The Hemodialysis Novel Therapies Consortium – Gut Microbiome and p-Inulin in Hemodialysis study is funded by the NIDDK.

#### **DSMB RESPONSIBILITIES**

The initial responsibility of the DSMB will be to review the study protocols, consent documents and plans for data safety monitoring, and approve the initiation of these clinical trials. After this approval, and at periodic intervals during the course of the trials, the DSMB responsibilities are to:

- review and approve major changes in the research protocol, informed consent documents and plans for data safety and monitoring, including all proposed revisions;
- evaluate the progress of the trial, including periodic assessments of data quality and timeliness, participant recruitment, accrual and retention, participant risk versus benefit, performance of the trial sites, and other factors that may affect study outcome;
- consider factors external to the study when relevant information becomes available, such as scientific or therapeutic developments that may have an impact on the safety of the participants or the ethics of the trial;
- protect the safety of the study participants;
- report on the safety and progress of the trial;
- make recommendations to the NIDDK, the Steering Committee and, if required, to the Food and Drug Administration (FDA) and the Institution Review Boards (IRBs) concerning continuation, termination or other modifications of the trial based on the observed beneficial or adverse effects of the treatment under study;
- if appropriate, conduct interim analysis of efficacy in accordance with stopping rules which are clearly defined in advance of data analysis and have the approval of the DSMB;
- ensure the confidentiality of the trial data and the results of monitoring;
- assist the NIDDK by commenting on any problems related to study conduct, enrollment, sample size, and/or data collection.

#### **MEMBERSHIP**

The DSMB will consist of at least eight members. Five participating members will constitute a quorum. The members have been appointed by the NIDDK. Members of the DSMB shall have no financial, scientific, or other conflict of interest with the studies. Collaborators or associates of the investigators in this trial are not eligible to serve on the DSMB. Written documentation attesting to absence of conflict of interest is required.

Dr. Paul Palevsky of University of Pittsburgh School of Medicine has been selected by the NIDDK to serve as the DSMB Chairperson for the remainder of the study. He is responsible for overseeing the meetings and developing the agenda in consultation with the NIDDK Program Directors, Dr. Paul Kimmel and Dr. John Kusek. Dr. Kimmel will serve as the DSMB Executive Secretary. The Chairperson is the contact

person for the DSMB. Other NIDDK official (s) or NIDDK appointee (s) may serve as an ex-officio member (s) of the DSMB. The DCC, University of Pennsylvania, shall provide the logistical management for the DSMB, in coordination with NIDDK (Dr. Yining Xie, as point of contact). Whenever possible, Dr. Robert Star, Director of the Division of Kidney, Urology and Hematology of NIDDK will also attend meetings.

#### **BOARD PROCESS**

The DSMB will meet a minimum of once a year at the call of the Chair, with advance approval of the NIDDK Program Director. An NIDDK representative will be present at every meeting.

Meetings shall be closed to the public because discussions may address confidential patient data. Meetings are attended, when appropriate, by the principal investigator and members of his/her staff. Meetings may be convened as conference calls/webinars as well as in person. An emergency meeting of the DSMB may be called at any time by the Chairperson or by the NIDDK Program Director should questions of patient safety arise. The DSMB Chairperson should contact the NIDDK Program Director prior to convening the meeting.

#### MEETING FORMAT

An appropriate format for DSMB meetings consists of open, closed and executive sessions. This format may be modified as needed. A brief closed and/or an executive session will usually be held before the open session.

#### **Open Session:**

The members of the DSMB, the NIDDK staff, the steering committee, including the study biostatistician will attend the open session. Issues discussed will include the conduct and progress of the study, including patient recruitment, data quality, general adherence and toxicity issues, compliance with protocol, and any other logistical matters that may affect either the conduct or outcome of the study. Protocol amendments may also be presented in this session.

#### **Closed Session:**

The closed session will be attended by voting DSMB members, representatives from the NIDDK, or its appointees, and the study biostatistician. **The discussion at the closed session is completely confidential.** 

Analyses of <u>blinded</u> outcome data are reviewed by masked intervention groups, including baseline characteristics, primary and secondary outcomes, adverse events, adherence and dropouts, and examination of any relevant subgroups. However, the DSMB may request unmasking of the data for either safety or efficacy concerns.

# **Executive Session:**

The executive session will be attended by voting DSMB members, and the NIDDK Staff, or its appointees.

The DSMB will discuss information presented to it during the closed and open sessions and decide whether to recommend continuation or termination, protocol modification or other changes to the

conduct of the study in the Executive Session. The DSMB can become unblinded if trends develop either for benefit or harm to the participants.

Should the DSMB decide to issue a termination recommendation, a full vote of the DSMB will be required. In the event of a split vote, majority vote will rule and a minority report should be appended. Reasons for early termination may include:

- Serious adverse effects in the entire intervention group or in a dominating subgroup;
- Greater than expected beneficial effects;
- A statistically significant difference by the end of the study is improbable;
- Logistical or data quality problems so severe that correction is not feasible.

## **Final Open Session (optional):**

The final session may be attended by voting DSMB members, steering committee members, the study biostatistician or other study members, and the NIDDK staff.

The Chairperson of the DSMB or the NIDDK Staff shall report on the recommendations of the DSMB regarding study continuation and concerns regarding the conduct of the study. Requests regarding data presentation for subsequent meetings will be made. Scheduling of the next DSMB meeting may be discussed.

#### **REPORTS**

**Interim Reports**: Interim reports will be prepared by the Data Coordinating Center, located at the University of Pennsylvania. The reports will be distributed to the DSMB and the NIDDK Program Director at least 7 days prior to a scheduled meeting. These interim reports are numbered and provided in sealed envelopes within an express mailing package or by secure email as the DSMB prefers. The contents of the report are determined by the DSMB. Additions and other modifications to these reports may be directed by the DSMB on a one-time or continuing basis. Interim data reports generally consist of two parts:

Part 1 (**Open Session Report**) provides information on study aspects such as accrual, baseline characteristics, and other general information on study status. This report is generally shared with all investigators involved with the clinical trial. The reports contained in this section may include:

- o Comparison of Target Enrollment to Actual Enrollment by Month
- o Comparison of Target Enrollment to Actual Enrollment by Site
- Overall Subject Status by Site, including: Subjects Screened, Enrolled, Active, Completed and Terminated
- o Demographic and Key Baseline Characteristics by Group
- o Treatment Duration for Subjects who Discontinue Therapy
- o Adverse Events/Serious Adverse Events by Site and Subject

Part 2 (**Closed Session Report**) may contain data on study outcomes, including safety data, including serious adverse events or termination. Data will be presented by masked treatment groups; however, the DSMB may request that the treatment groups be unmasked to ensure that there are no untoward treatment effects. This report should not be viewed by any members of the clinical trial except the designated study statistician.

**Reports from the DSMB:** A formal report containing the recommendations for continuation or modifications of the study, prepared by the Executive Secretary with concurrence of the DSMB, will be sent to the Chair of the Steering Committee and the DCC PI. This report will also contain any recommendations of the NIDDK in reference to the DSMB recommendations. It is the responsibility of the DCC PI to distribute this report to all other PIs and to assure that copies are submitted to all the IRBs associated with the study.

Each report should conclude with a recommendation to continue or to terminate the study. This recommendation should be made by formal majority vote. A termination recommendation may be made by the DSMB at any time by majority vote. The NIDDK is responsible for notifying the Chair of the Steering Committee of a decision to terminate the study. In the event of a split vote in favor of continuation, a minority report should be contained within the regular DSMB report. The report should not include unblinded data, discussion of the unblinded data, or any other confidential data.

**Mailings to the DSMB:** On a scheduled basis, (as agreed upon by the DSMB) blinded safety data should be communicated to all DSMB members and the NIDDK Program Director. Any concerns noted by the DSMB should be brought to the attention of the NIDDK Program Director.

Access to Interim Data: Access to the accumulating endpoint data should be limited to as small a group as possible. Limiting the access to interim data to the DSMB members relieves the investigator of the burden of deciding whether it is ethical to continue to randomize patients and helps protect the study from bias in patient entry and/or evaluation.

#### CONFIDENTIALITY

All materials, discussions and proceedings of the DSMB are completely confidential. Members and other participants in DSMB meetings are expected to maintain confidentiality.